CLINICAL TRIAL: NCT03450993
Title: A SMART Approach to Reducing Atrial Fibrillation Symptoms
Brief Title: SMART Program for Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michelle Dossett, MD, PhD, MPH, Assistant Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018P000015
Record Dates: First submitted 2018-02-16; First posted 2018-03-01 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Paroxysmal Atrial Fibrillation; Stress
Keywords: Mind-Body
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate SMART Program Intervention (Experimental): Subjects will receive the SMART-3RP intervention following study enrollment.
  Interventions: Other: SMART Program
- Delayed SMART Program Intervention (Other): Subjects will record symptoms following enrollment and receive the SMART-3RP intervention approximately 3 months following study enrollment.
  Interventions: Other: SMART Program

INTERVENTIONS:
Other: SMART Program — This is an 8-week, multimodal resiliency program that targets stress with 4 main components: mind-body skills (participants learn a variety of meditation techniques, mini relaxations, walking meditation, and yoga), traditional stress management techniques, healthy lifestyle behaviors (sleep, exercise, nutrition, and social support), and cognitive reappraisal and adaptive coping skills (borrowed from cognitive behavioral therapy, acceptance and commitment therapy, and positive psychology)
  Other Names: Stress Management and Resiliency Training Relaxation Response Resiliency Program (SMART-3RP) or Stress Management and Resiliency Training Program (SMART Program)

SUMMARY:
This is a pilot study to test the effects of the SMART-3RP (Stress Management and Resiliency Training Relaxation Response Resiliency Program) on quality of life, mental health, arrhythmia burden, and heart rate variability (HRV) in patients with paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
Mind-body practices that elicit the relaxation response (RR) have been used worldwide to prevent and treat disease. The Stress Management and Resiliency Training - Relaxation Response Resiliency Program (SMART-3RP) is an 8-week manualized psycho-educational program that incorporates RR methods such as meditation or seated yoga along with cognitive skills building and lifestyle approaches to increase resiliency to stress. This study will use a randomized, wait-list controlled trial design to test the effects of the SMART-3RP on quality of life (QoL), mental health, arrhythmia burden, and HRV in patients with PAF. The program will be delivered virtually (via computer video conferencing), questionnaires will be completed, and physiological data as well as blood will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with documented recurrent symptomatic PAF.
* Currently on stable medical therapy for AF and willing to continue on the same treatment regimen while participating in the study.
* No current daily practice of yoga, meditation, guided imagery or other techniques that elicit the RR.
* Able to provide informed consent and to understand written and spoken English.

Exclusion Criteria:

* Allergy to adhesives that prevents wearing the HRV monitor.
* Patients unable or unwilling to participate in an intervention delivered via video conferencing.
* End Stage renal failure or heart failure, severe unstable medical or psychiatric disease.
* Patients deemed unable to complete protocol due to cognitive or other reasons.
* Patients on psychoactive medications will have eligibility determined by the PI or MD co-investigator on a case-by-case basis, and will be admitted to the study if medication is deemed stable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptoms as measured by the generalized anxiety disorder 7 item questionnaire (GAD-7). | Approximately 3 months (beginning of study to completion of the program)
Change in AF-related quality of life as measured by the Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT). | Approximately 3 months (beginning of study to completion of the program)
Change in depressive symptoms as measured by the Patient Health Questionnaire 8 item instrument (PHQ-8). | Approximately 3 months (beginning of study to completion of the program)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dossett, MD, PhD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States